CLINICAL TRIAL: NCT06139380
Title: Intranasal Ketamine Effectiveness in Reducing Intramuscular Injection Pain Before Sedation Among Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hadi Mirfazaelian, Assistant Professor of Emergency Medicine, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9911307010
Record Dates: First submitted 2023-11-06; First posted 2023-11-18 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Pain; Intranasal Ketamine
MeSH Terms: conditions — Pain | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: 2-group parallel double blind randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: We will blind medication administrator, care provider, and assessor in addition to the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intranasal ketamine (Active Comparator)
  Interventions: Drug: Ketamine
- Intranasal sterile water (Placebo Comparator)
  Interventions: Drug: Sterile water

INTERVENTIONS:
Drug: Ketamine — This is medication which is commonly used for sedation in the emergency department. At the analgesic dose, this medication can be used to reduce the pain via other routes such as intranasal.
  Arms: Intranasal ketamine
Drug: Sterile water — Intranasal sterile water was administered via syringe.
  Arms: Intranasal sterile water

SUMMARY:
Hypothesis: Intranasal administration of ketamine would reduce the intramuscular pain of ketamine injection in children who undergo procedural sedation and analgesia in the emergency department.

DETAILED DESCRIPTION:
Ketamine is a well-known medication in children's procedural sedation and analgesia. While it provides good analgesia along with sedation, its injection is painful and causes distress in children. Intranasal administration of Ketamine would reduce the intramuscular pain of ketamine injection in children who undergo procedural sedation and analgesia in the emergency department. This will also assess if intranasal administration would affect the depth of sedation and hospital length of stay of this group of patients.

ELIGIBILITY:
Inclusion Criteria:

• Children who need to undergo procedural sedation and analgesia

Exclusion Criteria:

* Weight over 33 Kg
* No Consent from parents/patient
* Needs immediate procedure due to patient's condition
* Growth/mental retardation
* Sensory deficit at the site of intramuscular injection

Ages: 12 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2023-12-02 (Actual); Primary Completion 2024-04-28 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Intramuscular injection pain | immediately after Intramuscular injection
  This will be assessed at the time of injection using FLACC scale.

SECONDARY OUTCOMES:
Hospital stay duration | 1 hours on average
  This will be assessed using modified Ramsay's sedation scale.
Adverse effects | 1 hours on average
  This will be assessed using the standard definition of the adverse effects.

CONTACTS AND LOCATIONS:
Locations (1):
- IKHC, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No